CLINICAL TRIAL: NCT02787616
Title: Validation of Candidate Rosacea Genes By Targeted Interrogation of Alleles and Assessment of Rosacea Co-morbidities
Brief Title: Genetic Basis of Rosacea
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Other Study IDs: R15006
Record Dates: First submitted 2016-04-18; First posted 2016-06-01 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Rosacea Group
  Interventions: Genetic: buccal swab
- Non-Rosacea Group
  Interventions: Genetic: buccal swab

INTERVENTIONS:
Genetic: buccal swab — cheek swab for DNA sampling

SUMMARY:
Rosacea is a common disease characterized by inflammation and vascular abnormalities of the facial skin and ocular surface. The exact pathogenesis of papulopustular rosacea is not well understood and current methods to treat this disease are often unsatisfactory. The purpose of this study is to develop gene expression profiles of papulopustular rosacea compared to those of normal skin. The investigators hope to better understand the abnormal gene functions that might contribute to this condition. This understanding may lead to the development of additional and better treatments for rosacea.

ELIGIBILITY:
Eligibility Criteria for Rosacea Group:

Inclusion criteria for rosacea participants:

1. Clinical signs and symptoms of rosacea (papulopustular or erythrotelangiectatic subtypes) present at enrollment as determined by the investigator
2. All four grandparents of European descent
3. Fitzpatrick skin type I or II
4. Age 18 years or older

Exclusion criteria for rosacea participants:

1. Unable or unwilling to provide written informed consent
2. Concomitant facial or medical condition that obscures diagnosis of rosacea (such as malar erythema from lupus erythematosus)
3. Acne vulgaris
4. Unable or unwilling to provide peripheral blood sample (a few teaspoons)
5. Inability for investigator to verify rosacea diagnosis on clinical examination due to rosacea treatment(s) leading to complete lack of signs and symptoms (such prior laser treatments, systemic tetracycline usage, etc.)
6. Use of topical prescription medications or procedures to the face within one month of enrollment
7. Women who are pregnant or lactating

Eligibility Criteria for Non-Rosacea Group:

Inclusion criteria for control participants:

1. No history of rosacea
2. No clinical signs or symptoms of rosacea
3. No family history of rosacea
4. All four grandparents of European descent
5. Fitzpatrick skin type I or II
6. Age 18 years or older

Exclusion criteria for control participants:

1. Unable or unwilling to provide written informed consent
2. Acne vulgaris
3. Unable or unwilling to provide peripheral blood sample (a few teaspoons)
4. Women who are pregnant or lactating
5. Use of topical prescription medications or procedures to the face within one month of enrollment
6. Skin conditions that might interfere with interpretation of procedure results (at the discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 individuals will be enrolled, 150 with dermatologist verified rosacea and 150 without rosacea.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Targeted interrogation of alleles and assessment of rosacea co-morbidities. | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Dermatology, Redwood City, California, United States